CLINICAL TRIAL: NCT02212821
Title: Brain Mechanisms Underlying the Effect of the Motilin Receptor Agonist Erythromycin on Hunger in Normal Weight Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Erythromycin_v6
Record Dates: First submitted 2014-03-21; First posted 2014-08-08 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): intravenous infusion
  Interventions: Drug: Placebo
- Erythromycin (Experimental): intravenous infusion
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin
  Arms: Erythromycin
Drug: Placebo — physiological saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the role of erythromycin, a prokinetic agent, on hunger, and the brain mechanism lying behind it.

ELIGIBILITY:
Inclusion Criteria:

* Female only.
* Age > 18 and < 60.
* Body Mass Index (BMI) of 19-25 kg/m2 (no weight change of more than 5 kg in the past three months).
* Not known to have any chronic medical illness or illnesses affecting the gastrointestinal, cardiovascular, or nervous systems, chronic pain or psychiatric disorder.
* If female not known to be pregnant.
* Not known to have any past upper gastrointestinal surgery.

Exclusion Criteria:

* Alcohol consumption > 7 drinks / week
* Major depression and chronic health conditions except controlled hypertension

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Functional brain images | 40 min after intervention
  The functional brain images will be taken via functional magnetic resonance imaging (fMRI), and be analysed via a software called SPM.

SECONDARY OUTCOMES:
hunger scores | every 10 minutes since the scan starts
  The hunger scores will be taken every 10 minutes since the scan starts via a 10 cm visual analogue scale.
gut hormones | every 10 min since the scan starts
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure gut hormones (motilin, ghrelin, CCK, PYY, GLP-1) by radioimmuno-assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — University of Leuven